CLINICAL TRIAL: NCT02396394
Title: Improving ART Retention and Adherence in Uganda: The WiseMama Study
Acronym: WiseMama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa J. Messersmith, Associate Professor, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-32876; 1R34MH103075-01A1 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: HIV
Keywords: HIV; ART Adherence; Retention in Care; Pregnant Women; Postpartum Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two-Step Adherence Feedback (Experimental): Intervention subjects will use an electronic pill container to hold their antiretroviral medications. Throughout the 6-month intervention (until subjects are 3 months post-partum), whenever an intervention subject fails to open her electronic pill container within 60 minutes of dose time (as indicated by lack of a pill container opening), she will be sent a text message reminder. Each intervention subject will also participate in monthly counseling sessions informed by the subject's most recent adherence data generated by the electronic pill container. The counselor will review the adherence report with the patient and 1) provide positive feedback when adherence is ≥95% in the previous month, or 2) discuss reasons for lapses and strategies for improving adherence when adherence is <95%.
  Interventions: Behavioral: Two-Step Adherence Feedback

INTERVENTIONS:
Behavioral: Two-Step Adherence Feedback — Intervention subjects will use an electronic pill container to hold their antiretroviral medications. Throughout the 6-month intervention (until subjects are 3 months post-partum), whenever an intervention subject fails to open her electronic pill container within 60 minutes of dose time (as indicated by lack of a pill container opening), she will be sent a text message reminder. Each intervention subject will also participate in monthly counseling sessions informed by the subject's most recent adherence data generated by the electronic pill container. The counselor will review the adherence report with the patient and 1) provide positive feedback when adherence is ≥95% in the previous month, or 2) discuss reasons for lapses and strategies for improving adherence when adherence is <95%.

SUMMARY:
WiseMama is designed to improve our understanding of interventions that are feasible and effective in helping HIV-positive pregnant and postpartum women to maintain high adherence to antiretroviral medications. The study will involve: a) assessing the feasibility and acceptability of the use of an innovative pill container equipped with real-time electronic data monitoring capacity by HIV positive pregnant and postpartum women in Uganda; b) generating preliminary effectiveness data of a 2-step feedback intervention on retention in care, antiretroviral therapy adherence, and clinical outcomes (CD4 and HIV viral load (VL)); c) exploring patient and provider perspectives on barriers and facilitators to retention in care and adherence to antiretroviral therapy in our study population.

DETAILED DESCRIPTION:
The investigators will implement WiseMama over 2.5 years by using a randomized controlled trial design to assess the 2-step feedback intervention. Researchers will also investigate barriers and facilitators to retention in care and antiretroviral therapy adherence using quantitative and qualitative research methods. 130 pregnant women will be enrolled in two (three if needed) clinic sites Uganda where "Option B+" is the standard of care. HIV-positive pregnant women enrolled in the study will be randomized to either an intervention or comparison group for the approximately 6-month intervention. The study will follow all women for an additional 3 months to determine the potential sustainability of the impact of the intervention. In addition to adherence and clinical data, quantitative and qualitative data will be collected using survey instruments, focus groups, and in-depth interviews. Analysis of these data will enable achievement of the specific aims and contribute to the scientific evidence base on effective approaches to promoting antiretroviral therapy adherence among pregnant and postpartum HIV positive women in Uganda and other similar populations in low-resource settings.

The specific aims of the study are to:

1. Test the acceptability and feasibility of the use of an electronic pill container by pregnant and postpartum women. Acceptability and feasibility of the device among pregnant and postpartum women in Uganda through the implementation of a randomized controlled trial (RCT, see specific aim 2).
2. Evaluate preliminary effectiveness of 2-step feedback on retention in care and ART adherence, and clinical outcomes of pregnant and postpartum women. We will evaluate preliminary effectiveness of the intervention by conducting a RCT.
3. Explore patient and provider perspectives on barriers and facilitators to retention in care and adherence to ART. We will use a mixed methods research approach to collect data from pregnant and postpartum women, health care providers, and counselors to elicit in-depth information regarding the behavioral, health systems-related, community, and social factors that influence adherence and retention in care.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive pregnant women
* Who are 18 years of age and above
* Who receive antenatal care, are ART-naive, and initiate ART at one of study sites in Central Uganda
* Pregnant women must be between 18 and 26 weeks of estimated gestation
* Be able to use a cell phone that can receive text messages
* Provide written informed consent.

Exclusion Criteria:

* Women who have had any previous experience with ARV medications, who cannot receive text messages in the home, or who are unwilling to provide written informed consent will not be allowed to participate

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of subjects who achieve >/= 95% adherence | Month 6 and Month 9
  Subjects will participate in the 6-month real-time feedback intervention using electronic pill container/device and data-informed counseling. Comparison patients will continue to be monitored by electronic pill container, but they will remain blinded to the adherence information generated by the devices, as will their counselors. The 6-month period will be followed by passive monitoring for 3 months.

SECONDARY OUTCOMES:
Proportion of subjects who achieve >/= 95% cumulative adherence over entire 6 months of intervention period | Month 6 and Month 9 of intervention
  Subjects will participate in the 6-month real-time feedback intervention using electronic pill container/device and data-informed counseling. Comparison patients will continue to be monitored by electronic pill container, but they will remain blinded to the adherence information generated by the devices, as will their counselors. The 6-month period will be followed by passive monitoring for 3 months.
Difference in proportion of subjects who achieve: a) attend all scheduled visits; b) collect ART medications pre- and post-delivery; and c) give birth at clinic site | Month 10
Difference in mean change in CD4 count between Months 0 and 7 (baseline/pre-intervention and post-intervention) in each study arm, measured as cells/µl. | Before intervention and at Month 6 (end of intervention)
Difference in % undetectable viral load (UDVL) (using a lower limit of detection of 50 copies/mL of HIV plasma) in Month 7 (post-intervention) in each study arm. | At enrollment and Month 7 (post-intervention)

OTHER OUTCOMES:
Proportion of subjects who report using device is convenient/easy | After Month 1 of intervention
  Feasibility and acceptability of electronic pill container

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Messersmith, PhD, MPH, Principal Investigator — Boston University Center for Global Health and Development
Locations (1):
- Mildmay Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sabin LL, Simmons E, Halim N, Hamer DH, Gifford AL, West RL, Larson A, Bonawitz R, Aroda P, Banigbe B, Holderman AJ, Murray L, DeSilva MB, Gasuza J, Mukasa B, Messersmith LJ. Real-time Feedback to Improve HIV Treatment Adherence in Pregnant and Postpartum Women in Uganda: A Randomized Controlled Trial. AIDS Behav. 2022 Dec;26(12):3834-3847. doi: 10.1007/s10461-022-03712-7. Epub 2022 Jun 15. PMID 35704124